CLINICAL TRIAL: NCT03313479
Title: Comparative Study of the Effect of Three Different Analgesic Techniques on the Incidence of Postoperative Nausea and Vomiting After Scleral Buckling Under General Anesthesia
Brief Title: the Effect of Three Different Analgesic Techniques on the Incidence of Postoperative Nausea and Vomiting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer of anesthesia, Cairo University
Other Study IDs: badawy 1
Record Dates: First submitted 2017-10-07; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Post Operative Nausea and Vomiting
Keywords: Nausea, vomiting
MeSH Terms: conditions — Vomiting; Nausea | interventions — Dexmedetomidine; Scleral Buckling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: GA and Dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- group 2: GA and peribulbar
- group3: GA and xylocaine gel

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be given with GS
  Other Names: Dexmedetomidine with scleral buckling
  Groups: Group 1

SUMMARY:
Postoperative nausea and vomiting (PONV) is a distressing adverse effect that may result in postoperative complications including bleeding, wound dehiscence, aspiration pneumonitis, as well as fluid and electrolyte imbalances Incidence of PONV after general anesthesia is about 30% in all post-surgical patients but up to 80% in high-risk patients despite advances in anesthetics and anesthesia techniques

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a distressing adverse effect that may result in postoperative complications including bleeding, wound dehiscence, aspiration pneumonitis, as well as fluid and electrolyte imbalances.

The incidence of PONV after general anesthesia is about 30% in all post-surgical patients but up to 80% in high-risk patients despite advances in anesthetics and anesthesia techniques.

Despite new antiemetic drugs the overall incidences remain high especially in subjects with increased patient-related risk-factors such as in female gender, non-smoking status, a history of motion sickness or previous PONV, inhalational anesthetics, certain types of surgery, and opioid use. Scleral buckling (SB) which is still thought to be the most efficacious and cost-effective primary procedure for the treatment of uncomplicated retinal detachment is often associated with postoperative pain as well as nausea and vomiting. Preoperative injections of local anesthetics via retrobulbar, peribulbar, or subtenon routes in patients undergoing vitreoretinal surgery under general anesthesia (GA) have been reported to reduce postoperative pain, nausea, and vomiting.

Topical lidocaine drops have also has been used intraoperatively to decrease the incidence and severity of the OCR and to prevent pain and PONV after strabismus surgery and vitrectomy without scleral buckling .

The current study was designed to compare the effect of three different analgesic techniques ; IV analgesia , peribulbar block and topical xylocaine jel on the incidence of ponv after scleral buckling under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* males or females
* aged between 18-80 years
* ASA physical status Ι&II -indicated for repair of retinal detachment with scleral buckling. -

Exclusion Criteria:

* Patients with cardiac, liver and/or kidney diseases
* coagulation defects or receiving anticoagulants
* hypersensitivity to the used drugs
* history of motion sickness or PONV
* diabetes mellitus
* gastrointestinal disease
* smokers
* menstruating ladies
* ASA status more than II

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergo repair of retinal detachment with scleral buckling
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-10-30 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
PONV | 8 hours post operative
  incidence of post operative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No